CLINICAL TRIAL: NCT01995279
Title: The Effects of a Single Session of Ear Acupuncture in Pain Sensation and Body Balance
Brief Title: Ear Acupuncture Reducing Pain and Improving Balance
Acronym: EARPIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, Paulo Barbosa de Freitas Junior, Associate Professor, Universidade Cruzeiro do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCS_EA
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; French Auriculotherapy; postural control; balance; posture
MeSH Terms: conditions — Low Back Pain | interventions — Auriculotherapy; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- French ear acupuncture (Experimental): Application of single session of French ear acupuncture at specific points used to reduce low back pain.
  Interventions: Device: French ear acupuncture
- Sham Ultrasound (Placebo Comparator): Sham ultrasound will be applied at lumbar spine.
  Interventions: Other: Sham Ultrasound

INTERVENTIONS:
Device: French ear acupuncture — Single session (20 minutes) of French ear acupuncture at specific location used to reduce low back pain.
  Other Names: Auriculotherapy
  Arms: French ear acupuncture
Other: Sham Ultrasound — Ultrasound turned off.
  Other Names: Ultrasound
  Arms: Sham Ultrasound

SUMMARY:
The aim of the present project is to examine the effects of single session of French ear acupuncture on pain sensation and on postural control in individuals with chronic low back pain.

We hypothesize that:

I) The application of French ear acupuncture at specific points to reduce low back pain would decrease pain intensity in patients with chronic low back pain.

II) The pain reduction would be greater for those individuals with low back pain who receive application of French ear acupuncture at specific points to reduce low back pain compared with patients who receive placebo treatment.

III) The application of French ear acupuncture at specific points to reduce back pain will have positive effect on the performance of the postural control system.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of back pain lasting more than 12 weeks
* Pain referred larger than 4 according to the 11-points pain scale

Exclusion Criteria:

* No other musculoskeletal injury,
* Individuals diagnosed with structural damage
* Individuals who performed a spine surgery
* Individuals who have sensory abnormalities or dizziness.
* Individuals may not be in physical therapy for reducing low back pain.
* Painkillers or anti-inflammatories use 24 hours before the experimental procedure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
11-point Short Pain Scale (SPS-11) | 20 minute
  Treatment: single session of French ear acupuncture. Placebo: 20 minute application of sham ultrasound

SECONDARY OUTCOMES:
Center of pressure sway area | 20 minute
  Treatment: single session of French ear acupuncture. Placebo: 20 minute application of sham ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Paulo B de Freitas, PhD, Principal Investigator — Associate Professor, Universidade Cruzeiro do Sul
Locations (1):
- Laboratório de Análise do Movimento, Universidade Cruzeiro do Sul, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ushinohama A, Cunha BP, Costa LO, Barela AM, Freitas PB. Effect of a single session of ear acupuncture on pain intensity and postural control in individuals with chronic low back pain: a randomized controlled trial. Braz J Phys Ther. 2016 Jul-Aug;20(4):328-35. doi: 10.1590/bjpt-rbf.2014.0158. Epub 2016 Jun 16. PMID 27556389